CLINICAL TRIAL: NCT03752476
Title: Impact of Number of Rank of B-lactam Antibiotics on Emergence on Multidrug Resistant Bacteria
Acronym: INOR Blact
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Estelle Dossot, Internal, Centre Hospitalier Universitaire de Besancon
Other Study IDs: Dossot
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2018-11-26 (Actual); Status verified 2018-11

CONDITIONS: Resistant Infection; Antibiotic Resistant Infection; Beta Lactam Resistant Bacterial Infection; Bacterial Resistance
Keywords: antibiotic resistant; multidrug resistant; Beta lactam

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- case: Patients are colonized patient by antimicrobial bacteria hospitalized in intensive care during the fist hospitalization in intensive care during 2016-2017.
  Interventions: Procedure: number of Beta lactam class prescription for the same infection
- control: Patients aren't colonized patient by antimicrobial bacteria hospitalized in intensive care during the fist hospitalization in intensive care during 2016-2017.
  Interventions: Procedure: number of Beta lactam class prescription for the same infection

INTERVENTIONS:
Procedure: number of Beta lactam class prescription for the same infection — Each number of Beta lactam prescription without interruption are compared

SUMMARY:
This study evaluates the impact of rank of Beta lactam antibiotics on emergence of mutlidrug resistant bacteria colonization in intensive care

It's retrospective case controle study. Cases are colonized patient by multidrug resistant bacteria hospitalized in intensive care during the fist hospitalization in intensive care. Temoin are patients with the same characteristics than case but no colonized by multidrug resistant bacteria.

DETAILED DESCRIPTION:
The emergence of multidrug resistant is a wordwide problem. B lactam resistant increase. The antibiotic prescription impact this problem.

B lactam antibiotic is prescribed everyday in intensive care unit. The switch of antibiotic is common. Antibiotic classes inclue a lot of rank with different spectum that impact the occurrence of resistant.

ELIGIBILITY:
Inclusion Criteria:

* all patient hospitalized more than 48 hours in intensive care unit in Besançon between january 2016 and december 2017

Exclusion Criteria:

* patient under guardianship
* patient allergic to Beta lactam
* colonization with mutidrug resistant the first week of hospitalization in intensive care unit

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all patient hospitalized more than 48 hours in intensive care unit in Besançon between january 2016 and december 2017
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
number of Beta lactam class prescription | 3 months

IPD SHARING:
Plan to Share IPD: No